CLINICAL TRIAL: NCT02252276
Title: Effects of Manual Therapy and Exercise in the Treatment of Recurrent Ankle Sprains: Randomised Trial
Brief Title: Effects of Manual Therapy and Exercise in the Treatment of Ankle Sprains
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Prof. Dr. Daniel Pecos Martín, Dr Daniel Pecos Martín, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M2013/031/20131120
Record Dates: First submitted 2014-09-23; First posted 2014-09-30 (Estimated); Last update posted 2014-09-30 (Estimated); Status verified 2014-09

CONDITIONS: Ankle Sprains
Keywords: Manual therapy; proprioception; exercises; ankle sprain
MeSH Terms: conditions — Ankle Injuries; Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental (Experimental): performed the same exercises and manual therapy during 4 weeks
  Interventions: Procedure: Experimental (proprioception exercises, muscle strengthening, joint mobilization)
- Control (Active Comparator): performed proprioceptive and strengthening exercises during 4 weeks
  Interventions: Procedure: Control (proprioception exercises, muscle strengthening)

INTERVENTIONS:
Procedure: Experimental (proprioception exercises, muscle strengthening, joint mobilization) — The experimental group performed a combined protocol of proprioception (the patient doing exercises standing on an unstable plane)exercises and muscle strengthening (The patient performed eccentric exercises to work the movement inversion of ankle), and joint mobilization techniques of the ankle joint two session per week, during four weeks
  Arms: Experimental
Procedure: Control (proprioception exercises, muscle strengthening) — The control group performed only proprioception exercises (the patient doing exercises standing on an unstable plane) and muscle strengthening (The patient performed eccentric exercises to work the movement inversion of ankle). Two sessión per week during four weeks
  Arms: Control

SUMMARY:
Objectives: To analyze the effects of proprioceptive and strengthening exercises versus the same exercises and manual therapy on the recurrent ankle sprain management.

Design: A randomized clinical trial with two intervention groups and triple blind.

Settings: University Hospital.

Participants: Fifty-four patients with previous history of recurrent ankle sprains, regular sports practice and pain during the physical activity, randomly assigned to experimental or control group.

Intervention: Control group performed 4 weeks of proprioceptive and strengthening exercises; experimental group performed 4 weeks of the same exercises combined with manual therapy.

Main Outcomes Measures: Pain, ankle instability, pressure pain threshold (PPT), ankle eversion strength, and active range of motion in ankle joint. The measures were taken before, after and one month after the interventions.

DETAILED DESCRIPTION:
The recurrent ankle sprain means the most frequent complication from the ankle sprain and the previous phase of the chronic ankle stability (CAI), which involves between 20 - 41% of all ankle sprains.

Residual pain concerns the first symptom after instability in most of the cases, but patients also show reduced ankle joint position sense, ankle range of motion, and strength of ankle inversion muscles.

Proprioception exercises on multiplane and unstable platforms, as well as strengthening through eccentric exercises report benefits in pain and function, suggesting the active therapy as the most effective treatment instead of passive manual therapy in chronic phases.

However, several studies analyzed the effects of the manual therapy in the management of the ankle sprain recurrence: the posterior gliding of astragalus and the tibiotarsal joint coaptation improved the ankle range of motion, which was related with recurrent ankle sprain and its residual symptoms.

Despite the benefits from active and passive therapy, very few authors up to date investigated the combination of both clinical approach in the recurrent ankle sprain. Literature analyzed the effects of a combined program including exercises to the manual therapy in acute ankle sprain and concluded that the variety in the manual therapy techniques reported more pain release and improved function.

Besides, based on the effects of joint mobilization techniques, the neurodynamic mobilization could be an appropriate therapy, due to the neural distribution of fibular nerve through the ankle joint, but no studies to date to our knowledge included this technique as part of the recurrent ankle sprain management.

This study aimed to analyze the effects of proprioceptive and strengthening exercises versus the same exercises and manual therapy on the recurrent ankle sprain management.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with previous history of recurrent ankle sprain

Exclusion Criteria:

* Subjects with surgical treatment, previous fractures on lower limb and/or adjacent pathologies were excluded from the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2014-01; Primary Completion 2014-04 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Pain | Change from baseline at one month
  All the subjects showed their pain level from 0 (no pain) to 10 (maximum pain) in a Visual Analogical Scale (VAS).

SECONDARY OUTCOMES:
The Cumberland Ankle Instability Tool (CAIT) | Change from baseline at one month
Pressure Pain Threshold (PPT) | Change from baseline at one month
  An algometer Wagner FPI 10-WA was used to determine the PPT in the anterior talofibular ligament, the calcaneofibular ligament, tibial malleolus, and fibular malleolus. The pressure was perpendicular hold in each structure, while patients were positioned sidelined on the unaffected side with knee and hip semiflexion
Active range of motion in ankle joint | Change from baseline at one month
  A standard goniometer was employed. Patients were seated in 90º knee flexion and ankle neutral position. The goniometer fulcrum was placed over the lateral malleolus, with its proximal arm over the fibular diaphysis and distal arm over the fifth metatarsal. Patients were asked to actively perform a flexion and extension of ankle.
Strength in ankle flexion and extension | Change from baseline at one month
  dynamic dynamometry with MicroFet-2 was used while patients were positioned in supine and lower limb on the therapeutic table. From this position, patients performed ankle flexion and extension. The test-retest reliability of this tool has been previously shown

CONTACTS AND LOCATIONS:
Overall Officials: Tomas Gallego-Izquierdo, Dr, Principal Investigator — Alcala University
Locations (1):
- Alcalá University, Alcalá de Henares, Madrid, Spain